CLINICAL TRIAL: NCT00024544
Title: A Phase I/II, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Pilot Study of SB 240683 in Patients With Symptomatic Steroid-Naive Asthma
Brief Title: Pilot Study in Patients With Symptomatic Steroid-Naive Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Facet Biotech (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 683-803
Record Dates: First submitted 2001-09-19; First posted 2001-09-20 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2012-03

CONDITIONS: Asthma
Keywords: asthma; anti-IL-4 monoclonal antibody; pascolizumab
MeSH Terms: conditions — Asthma

INTERVENTIONS:
Drug: anti-IL-4 monoclonal antibody (pascolizumab)

SUMMARY:
The purpose of the study is to evaluate an investigational medication to treat chronic asthma. The research is being conducted at 20 clinical research sites in the US and is open to both men and women ages 18 to 70 years. Participants in the study will have a number of visits to a research site over an 8-month period. All study-related care and medication is provided to qualified participants at no cost. This includes all visits, examinations and laboratory work.

ELIGIBILITY:
Inclusion Criteria:

* At least a 6-month history of asthma
* No use of inhaled, oral or injectable steroids for at least 1 month prior to enrollment

Exclusion Criteria:

* Patients with > 10 pack years of smoking history or smoking within 12 months of study enrollment
* No significant disease other than asthma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120
Dates: Start 2001-08; Primary Completion 2003-02 (Actual); Study Completion 2003-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - Allergy Research Foundation, Los Angeles, California
  - Southern California Research, Mission Viejo, California
  - Clinical Trials of Orange Cnty., Inc., Orange, California
  - Allergy Associates Medical Group, Inc., San Diego, California
  - Allergy and Asthma Associates Santa Clara Valley Research Center, San Jose, California
  - Bensch Research Associates, Stockton, California
  - National Jewish Medical and Research Center, Denver, Colorado
  - ICSL Clinical Studies, Normal, Illinois
  - Respiratory Therapy and Pulmonary Clinical Research Brigham & Women's Hospital, Boston, Massachusetts
  - New England Clinical Studies, North Dartmouth, Massachusetts
  - Clinical Research Institute, Minneapolis, Minnesota
  - The Clinical Research Center, LLC, St Louis, Missouri
  - Center for Allergy, Asthma and Immunology, Creighton University, Omaha, Nebraska
  - Princeton Center for Clinical Research, Princeton, New Jersey
  - Allergy, Asthma, and Dermatology Research Center, LLC, Lake Oswego, Oregon
  - Valley Clinical Research Center, Easton, Pennsylvania
  - Clinical Trials North Houston, Houston, Texas
  - University of Wisconsin Medical School, Madison, Wisconsin